CLINICAL TRIAL: NCT02100813
Title: Safety and Efficacy of Escalating Doses of LEO 43204 Applied Once Daily for Two Consecutive Days on Full Balding Scalp in Subjects With Actinic Keratosis
Brief Title: Safety and Efficacy of Doses of LEO 43204 Once Daily for Two Consecutive Days on Full Balding Scalp in Subjects With Actinic Keratosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0084-1014; 2014-000037-23 (EudraCT Number)
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2018-11

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — LEO 43204

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1: LEO 43204 (Other): Open-label, dose escalation, 2 days treatment
  Interventions: Drug: LEO 43204
- Part 2: LEO 43204 x dose (Active Comparator): X dose for 2 days treatment
  Interventions: Drug: LEO 43204
- Part 2: LEO 43204 Y dose (Active Comparator): Y dose for 2 days treatment
  Interventions: Drug: LEO 43204
- Part 2: Placebo (Placebo Comparator): Placebo for 2 days treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEO 43204
  Arms: Part 1: LEO 43204; Part 2: LEO 43204 Y dose; Part 2: LEO 43204 x dose
Drug: Placebo
  Arms: Part 2: Placebo

SUMMARY:
To identify the Maximum Tolerated Dose levels of LEO 43204 after once daily treatment for two consecutive days and to evaluate efficacy of LEO 43204 in two doses after once daily treatment for two consecutive days compared to vehicle

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Subjects with 5 to 20 clinically typical, visible and discrete AKs on the full balding scalp.
* Part 2: Subjects with 5 to 20 clinically typical, visible and discrete AKs on the full balding scalp

Exclusion Criteria:

* Location of the treatment area

  * within 5 cm of an incompletely healed wound
  * within 5 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC)
* Prior treatment with ingenol mebutate gel on the treatment area
* Lesions in the treatment areas that have

  * atypical clinical appearance (e.g., hypertrophic, hyperkeratotic or cutaneous horns) and/or
  * recalcitrant disease (e.g., did not respond to cryotherapy on two previous occasions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Weiss, MD, Principal Investigator — Gwinnett Clinical Research Center, Inc.
Locations (1):
- Gwinnett Clinical Research Center, Inc., Snellville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 7 centres in the US into Part 1 of the trial. First participant was enrolled on 14-05-14 and the last subject´s last visit (LSLV) was on 12-08-14. Participants were recruited in 11 centres in the US and 5 centres in Germany into Part 2 of trial. First participant was enrolled on 03-09-14 and LSLV was on 02-03-14.
Groups:
- Part 1 - 0.018% Cohort: Part 1 - Dose escalation
  Once daily application with LEO 43204 gel (ingenol disoxate) 0.018% for two consecutive days on balding scalp.
- Part 1 - 0.025% Cohort: Part 1 - Dose escalation
  Once daily application with LEO 43204 gel 0.025% for two consecutive days on balding scalp.
- Part 1 - 0.037% Cohort: Part 1 - Dose escalation
  Once daily application with LEO 43204 gel 0.036% for two consecutive days on balding scalp.
- Part 1 - 0.05% Cohort: Part 1 - Dose escalation
  Once daily application with LEO 43204 gel 0.05% for two consecutive days on balding scalp.
- Part 1 - 0.075% Cohort: Part 1 - Dose escalation
  Once daily application with LEO 43204 gel 0.075% for two consecutive days on balding scalp.
- Part 2 - Vehicle: Part 2 - Dose finding
  Once daily application with LEO 43204 gel vehicle for two consecutive days on balding scalp.
- Part 2 - 0.037%: Part 2 - Dose finding
  Once daily application with LEO 43204 gel 0.037% for two consecutive days on balding scalp.
- Part 2 - 0.05%: Part 2 - Dose finding
  Once daily application with LEO 43204 gel 0.05% for two consecutive days on balding scalp.
Period: Overall Study
Arm/Group | Part 1 - 0.018% Cohort | Part 1 - 0.025% Cohort | Part 1 - 0.037% Cohort | Part 1 - 0.05% Cohort | Part 1 - 0.075% Cohort | Part 2 - Vehicle | Part 2 - 0.037% | Part 2 - 0.05%
Started | 10 | 11 | 12 | 12 | 12 | 32 | 64 | 67
Completed | 10 | 11 | 12 | 12 | 12 | 32 | 64 | 66
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1 - 0.018% Cohort: Part 1 - Dose escalation
  Once daily application with LEO 43204 gel 0.018% for two consecutive days on balding scalp.
- Part 1 - 0.037% Cohort: Part 1 - Dose escalation
  Once daily application with LEO 43204 gel 0.037% for two consecutive days on balding scalp.
- Total: Total of all reporting groups
Arm/Group | Part 1 - 0.018% Cohort | Part 1 - 0.025% Cohort | Part 1 - 0.037% Cohort | Part 1 - 0.05% Cohort | Part 1 - 0.075% Cohort | Part 2 - Vehicle | Part 2 - 0.037% | Part 2 - 0.05% | Total
Number analyzed (Participants) | 10 | 11 | 12 | 12 | 12 | 32 | 64 | 67 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 4 | 4 | 2 | 9 | 9 | 14 | 47
  >=65 years | 8 | 8 | 8 | 8 | 10 | 23 | 55 | 53 | 173
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 11 | 12 | 12 | 12 | 32 | 64 | 67 | 220
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 12 | 12 | 12 | 24 | 49 | 51 | 181
  Germany | 0 | 0 | 0 | 0 | 0 | 8 | 15 | 16 | 39

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants Experiencing a Dose-limiting Toxicity (DLT)
Description: The number participants experiencing a DLT was used to identify the maximum tolerated dose (MTD) of LEO 43204 after once daily treatment for 2 consecutive days.The MTD was defined as the highest dose level with less than 4 out of 12 participants experiencing a DLT.
  A DLT was defined as:
  * Erosion/ulceration Grade 4 on the Local Skin Response (LSR) scale
  * Other clinically relevant signs or symptoms observed, which the International Co-ordinating Investigator judges to be counted as a DLT.
  The Local Skin Responses consists of the following 6 categories: Erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration. Each individual LSR category are given a numeric grade of severity from 0-4. Grade 0 being no presence and Grade 4 being the highest grade of severity.
Time Frame: From Day 1 up to and including Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - 0.018% Cohort | Part 1 - 0.025% Cohort | Part 1 - 0.037% Cohort | Part 1 - 0.05% Cohort | Part 1 - 0.075% Cohort
Number analyzed (Participants) | 10 | 11 | 12 | 12 | 12
Participants
  Yes | 0 | 0 | 0 | 0 | 0
  No | 10 | 11 | 12 | 12 | 12

2. Primary Outcome: Part 2: Percent Reduction From Baseline in Actinic Keratosis (AK) Lesion Count
Description: Percent reduction from baseline in clinically visible actinic keratosis lesions (AKs) in the selected treatment area.
Time Frame: From baseline to Week 8
Measure: Mean (95% Confidence Interval); unit: percentage of reduction
Arm/Group | Part 2 - Vehicle | Part 2 - 0.037% | Part 2 - 0.05%
Number analyzed (Participants) | 32 | 64 | 67
percentage of reduction | 12.6 [-9.5 to 30.3] | 72.7 [66.9 to 77.5] | 78.5 [73.7 to 82.5]
Statistical Analysis 1: Comparison: Part 2 - Vehicle vs Part 2 - 0.037%; Negative binominal regression with log baseline count as offset variable and treatment group and analysis site as factors; Test type: Superiority or Other; p < 0.001, Negative binomial regression; Rate ratio = 0.31, 95% CI 2-sided [0.23 to 0.42]
Statistical Analysis 2: Comparison: Part 2 - Vehicle vs Part 2 - 0.05%; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Negative binomial regression; Rate ratio = 0.25, 95% CI 2-sided [0.18 to 0.33]
Statistical Analysis 3: Comparison: Part 2 - 0.037% vs Part 2 - 0.05%; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.096, Negative binomial regression; Rate ratio = 0.79, 95% CI 2-sided [0.59 to 1.04]

3. Secondary Outcome: Part 2: Participants With Complete Clearance of AKs
Description: Complete clearance of AKs at Week 8 was defined as a 100% reduction from baseline in AK count.
Time Frame: From baseline to Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 - Vehicle | Part 2 - 0.037% | Part 2 - 0.05%
Number analyzed (Participants) | 32 | 64 | 67
percentage of participants | 3.1 [0.1 to 16.2] | 21.9 [12.5 to 34] | 29.9 [19.3 to 42.3]
Statistical Analysis 1: Comparison: Part 2 - Vehicle vs Part 2 - 0.037%; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority or Other; p = 0.007, Log binomial regression; Ratio of clearance rates = 7.02, 95% CI 2-sided [1.53 to 124]
Statistical Analysis 2: Comparison: Part 2 - Vehicle vs Part 2 - 0.05%; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority or Other; p = 0.001, Log binomial regression; Ratio of clearance rates = 8.82, 95% CI 2-sided [1.99 to 154.5]
Statistical Analysis 3: Comparison: Part 2 - 0.037% vs Part 2 - 0.05%; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority or Other; p = 0.43, Log binomial regression; Ratio of clearance rates = 1.26, 95% CI 2-sided [0.72 to 2.31]

4. Secondary Outcome: Part 2: Participants With Partial Clearance of AKs
Description: Partial clearance of AKs at Week 8 was defined as at least 75% reduction from baseline in AK count.
Time Frame: From baseline to Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 - Vehicle | Part 2 - 0.037% | Part 2 - 0.05%
Number analyzed (Participants) | 32 | 64 | 67
percentage of participants | 6.3 [0.8 to 20.8] | 54.7 [41.7 to 67.2] | 59.7 [47.0 to 71.5]
Statistical Analysis 1: Comparison: Part 2 - Vehicle vs Part 2 - 0.037%; Test type: Superiority or Other; p < 0.001, Log binomial regression; Ratio of clearance rates = 8.73, 95% CI 2-sided [2.93 to 51.66]
Statistical Analysis 2: Comparison: Part 2 - Vehicle vs Part 2 - 0.05%; Test type: Superiority or Other; p < 0.001, Log binomial regression; Ratio of clearance rates = 9.55, 95% CI 2-sided [3.22 to 56.4]
Statistical Analysis 3: Comparison: Part 2 - 0.037% vs Part 2 - 0.05%; Test type: Superiority or Other; p = 0.55, Log binomial regression; Ratio of clearance rates = 1.09, 95% CI 2-sided [0.81 to 1.49]

ADVERSE EVENTS:
Time Frame: Part 1: From Day 1 to Week 2 Part 2: From Day 1 to Week 8
Groups:
- Part 1 - 0.025% Cohort: Part 1 - Dose escalation
  Once daily application with LEO 43204 gel 0.025%for two consecutive days on balding scalp.
Arm/Group | Part 1 - 0.018% Cohort | Part 1 - 0.025% Cohort | Part 1 - 0.037% Cohort | Part 1 - 0.05% Cohort | Part 1 - 0.075% Cohort | Part 2 - Vehicle | Part 2 - 0.037% | Part 2 - 0.05%
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/12 | 0/12 | 0/12 | 0/32 | 2/64 | 3/67
Other Adverse Events (participants affected / at risk) | 7/10 | 7/11 | 12/12 | 10/12 | 12/12 | 4/32 | 47/64 | 50/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - 0.018% Cohort (N=10) | Part 1 - 0.025% Cohort (N=11) | Part 1 - 0.037% Cohort (N=12) | Part 1 - 0.05% Cohort (N=12) | Part 1 - 0.075% Cohort (N=12) | Part 2 - Vehicle (N=32) | Part 2 - 0.037% (N=64) | Part 2 - 0.05% (N=67)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - 0.018% Cohort (N=10) | Part 1 - 0.025% Cohort (N=11) | Part 1 - 0.037% Cohort (N=12) | Part 1 - 0.05% Cohort (N=12) | Part 1 - 0.075% Cohort (N=12) | Part 2 - Vehicle (N=32) | Part 2 - 0.037% (N=64) | Part 2 - 0.05% (N=67)
Application site pruritus (General disorders) | 3 (3) | 3 (3) | 7 (7) | 5 (5) | 9 (10) | 1 (1) | 16 (18) | 18 (18)
Application site pain (General disorders) | 2 (3) | 4 (5) | 12 (18) | 9 (16) | 12 (17) | 2 (2) | 31 (42) | 38 (51)
Application site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Application site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Application site discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site hyperaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental exposure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Circumoral oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram u-wave abnormality (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 5 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visceral larva migrans (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.